CLINICAL TRIAL: NCT02131298
Title: A Phase 1, Open-Label, Fixed-Sequence 2-Period Study To Investigate The Effect Of Multiple Doses Of Itraconazole On The Single Dose Pharmacokinetics of Palbociclib (PD-0332991) In Healthy Volunteers
Brief Title: Effect Of Itraconazole On The Pharmacokinetics Of Palbociclib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481016
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Palbociclib; Itraconazole; Pharmacokinetics; Drug-Drug Interaction Study; Healthy Volunteers
MeSH Terms: interventions — palbociclib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fixed sequence (Other): Fixed sequence study with treatment A of palbociclib alone, followed by treatment B (palbociclib with itraconazole)
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib plus itraconazole

INTERVENTIONS:
Drug: Palbociclib Alone — A single 125 mg dose of palbociclib free base capsule given orally alone in the fed state, followed by 120 hours of PK sample collection
  Other Names: Palbociclib, PD-0332991
Drug: Palbociclib plus itraconazole — Itraconazole 200 mg once daily with food for a total of 11 days; on Day 5, a single oral 125 mg dose of palbociclib will be given with itraconazole after a meal, followed by 168 hours of PK sample collection.
  Other Names: Palbociclib (PD-0332991); Itraconazole (Sporanox)

SUMMARY:
This study is designed to evaluate the potential effect of itraconazole on the pharmacokinetics of palbociclib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Body mass index of 17.5 to 30.5 kg/m2, and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic diseases.
* Any condition possibly affecting drug absorption.
* A positive urine drug screen or alcohol breath test.
* Pregnant female subjects; breast feeding female subjects, female subjects of childbearing potential, male subjects with partners currently pregnant, male subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0 to 168 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0 to 168 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 to 168 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0 to 168 hours
Plasma Decay Half-Life (t1/2) | 0 to 168 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 0 to 168 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0 to 168 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481016&StudyName=Effect%20Of%20Itraconazole%20On%20The%20Pharmacokinetics%20Of%20Palbociclib